CLINICAL TRIAL: NCT04355442
Title: Evolution of Maxillofacial Trauma Activity During COVID-19 Containment Measures: a French Multicentric Comparative Observational Study
Brief Title: Evolution of Facial Trauma During COVID Containment Measures
Acronym: Traumax
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Unités de CMF des CHU de Paris (Dr Davrou - Pitié salpetrière) (Unknown); Amiens (Dr Dapke) (Unknown); Nantes (Pr Corre) (Unknown); Toulouse (Pr Lauwers - Purpan) (Unknown); Marseille (Dr Foletti - La conception) (Unknown); Nice (Dr Savoldelli) (Unknown); Clermont Ferrand (Dr Sesque) (Unknown); Perpignan (Dr Llobet) (Unknown); Lyon (Dr Bourlet - Croix Rousse) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0228
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-04

CONDITIONS: Maxillofacial Injuries; Skull Fractures; COVID-19
Keywords: Pandemics; Maxillofacial fractures; Facial trauma; Containment; Quarenteen; Outbreak
MeSH Terms: conditions — Maxillofacial Injuries; Skull Fractures; COVID-19 | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- contained patients: contained patients
  Interventions: Procedure: Facial fractures reduction or osteosynthesis
- Comparative patients: Comparative patients
  Interventions: Procedure: Facial fractures reduction or osteosynthesis

INTERVENTIONS:
Procedure: Facial fractures reduction or osteosynthesis — Facial fractures reduction or osteosynthesis

SUMMARY:
The COVID-19 global pandemic has led to a major professional and social national reorganization: professional because it involves a redeployment of medical staff and material resources, and social because it imposes prolonged containment measures on an entire population.

The maxillofacial trauma activity is mainly linked to sports or leisure accidents, fights and road accidents.

It seems to appear since the beginning of containment measures a significant drop in maxillofacial trauma activity at the national level, which, if it is demonstrated in a significant way in several French hospital centers, would allow to redeploy the material and human resources related to this activity on sectors in tension due to the pandemic.

DETAILED DESCRIPTION:
This study will compare maxillo-facial activity during the first month of COVID-19 containment measures in France with a comparable period in 2018 and 2019. This comparison will be made in 10 major French hospital centers.

ELIGIBILITY:
Inclusion criteria:

* Maxillo-facial fracture
* Requiring
* Trauma that occured between March 16 and April 15, 2020 or 2018 or 2019
* All ages

Exclusion criteria:

* Patients who refused the collection of their data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with facial trauma requiring surgery
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
evolution of number of maxillofacial trauma | 1 year
  evolution of number of maxillofacial trauma during COVID-19 first month of containment measures compared to the same period in 2018 and 2019.the number of patients from different investigator centers operated for a facial fracture occurring between March 16, 2020 and April 15, 2020 will be compared to the number of patients in these same centers operated for a facial fracture during the same period in 2018 and in 2019. A sub-group analysis, by center, will also be carried out.

SECONDARY OUTCOMES:
variability in terms of type of trauma | 1 year
  study of variability in terms of type of trauma with and without confinement.
Comparative assessment of types of trauma by the inter-regional variability | 1 year
  Comparative assessment of types of trauma by the inter-regional variability : study of the inter-regional variability of maxillofacial trauma

CONTACTS AND LOCATIONS:
Overall Officials: Marie de BOUTRAY, PH, Study Director — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC